CLINICAL TRIAL: NCT02175966
Title: Short Duration Combination Therapy With Daclatasvir, Asunaprevir, BMS-791325 and Sofosbuvir in Subjects Infected With Chronic Hepatitis C (FOURward Study)
Brief Title: Short Duration Combination Therapy With Daclatasvir, Asunaprevir, BMS-791325 and Sofosbuvir in Subjects Infected With Chronic Hepatitis-C (FOURward Study)
Acronym: FOURward
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI443-131
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: DCV/ASV/BMS-791325+Sofosbuvir (Experimental): Initial Therapy:
  Daclatasvir/Asunaprevir/BMS-791325 [30 mg (as the free base)/200 mg/75 mg (as the free base)] film coated Fixed Dose Combination tablet twice daily orally for 4 weeks
  Sofosbuvir 400 mg tablet once daily orally for 4 weeks
  Interventions: Drug: DCV/ASV/BMS-791325; Drug: Sofosbuvir
- Arm 2: DCV/ASV/BMS-791325 + Sofosbuvir (Experimental): Initial Therapy
  Daclatasvir/Asunaprevir/BMS-791325 [30 mg (as the free base)/200 mg/75 mg (as the free base)] film coated Fixed Dose Combination tablet twice daily orally for 6 weeks
  Sofosbuvir 400 mg tablet once daily orally for 6 weeks
  Interventions: Drug: DCV/ASV/BMS-791325; Drug: Sofosbuvir
- Rescue Therapy: Arm 1:DCV/ASV/BMS-791325+RBV±PegIFNα-2a (Experimental): Daclatasvir/Asunaprevir/BMS-791325 [30 mg (as the free base)/200 mg/75 mg (as the free base)] film coated Fixed Dose Combination tablet twice daily orally for 12 weeks
  Ribavirin 200 mg tablets twice daily (1000 or 1200 mg per day based on weight) orally for 12 weeks
  With or without Peginterferon α-2a 180 µg solution for injection subcutaneously once weekly for 12 weeks
  Interventions: Drug: DCV/ASV/BMS-791325; Drug: Ribavirin; Drug: Peginterferon α-2a
- Rescue Therapy: Arm 2: Sofosbuvir + RBV + PegIFNα-2a (Other): Sofosbuvir 400 mg tablet once daily orally for 12 weeks
  Ribavirin 200 mg tablets twice daily (1000 or 1200 mg per day based on weight) orally for 12 weeks
  Peginterferon α-2a 180 µg solution for injection subcutaneously once weekly for 12 weeks
  Interventions: Drug: Ribavirin; Drug: Sofosbuvir; Drug: Peginterferon α-2a

INTERVENTIONS:
Drug: DCV/ASV/BMS-791325
  Arms: Arm 1: DCV/ASV/BMS-791325+Sofosbuvir; Arm 2: DCV/ASV/BMS-791325 + Sofosbuvir; Rescue Therapy: Arm 1:DCV/ASV/BMS-791325+RBV±PegIFNα-2a
Drug: Ribavirin
  Arms: Rescue Therapy: Arm 1:DCV/ASV/BMS-791325+RBV±PegIFNα-2a; Rescue Therapy: Arm 2: Sofosbuvir + RBV + PegIFNα-2a
Drug: Sofosbuvir
  Other Names: Sovaldi®
  Arms: Arm 1: DCV/ASV/BMS-791325+Sofosbuvir; Arm 2: DCV/ASV/BMS-791325 + Sofosbuvir; Rescue Therapy: Arm 2: Sofosbuvir + RBV + PegIFNα-2a
Drug: Peginterferon α-2a
  Arms: Rescue Therapy: Arm 1:DCV/ASV/BMS-791325+RBV±PegIFNα-2a; Rescue Therapy: Arm 2: Sofosbuvir + RBV + PegIFNα-2a

SUMMARY:
The purpose of the study is to determine whether the combination of Daclatasvir (DCV), Asunaprevir (ASV), BMS-791325 and Sofosbuvir is effective and safe in treating Hepatitis-C virus.

DETAILED DESCRIPTION:
Allocation:

Initial Therapy: Randomized Controlled Trial: Participants are assigned to intervention groups by chance

Rescue Therapy: Nonrandomized Trial: Participants are expressly assigned to intervention groups through a non-random method such as physician choice

Number of Arms:

Initial Therapy: 2 Groups

Rescue Therapy: 2 Groups

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Males and Females ≥18 years of age, inclusive
* Chronic HCV infection Genotype 1 only
* Non-cirrhotic
* Treatment naive subjects with no previous exposure to an Interferon formulation (ie, IFNα, pegIFNα), ribavirin (RBV) or HCV Direct Acting Antiviral (DAA) (protease, polymerase inhibitor, etc.)

Exclusion Criteria:

* HCV Genotype other than Genotype 1
* Documented or suspected hepatocellular carcinoma
* Evidence of decompensated liver disease
* Contraindication(s) to Peg/RBV therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2015-01-28 (Actual); Study Completion 2015-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Inland Empire Liver Foundation, Rialto, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - Indiana University Health - University Hospital, Indianapolis, Indiana
  - Indiana University Med Center, Indianapolis, Indiana
  - Johns Hopkins University, Lutherville, Maryland
  - Texas Liver Institute, San Antonio, Texas

REFERENCES:
- [Derived] Sulkowski MS, Flamm S, Kayali Z, Lawitz EJ, Kwo P, McPhee F, Torbeyns A, Hughes EA, Swenson ES, Yin PD, Linaberry M. Short-duration treatment for chronic hepatitis C virus with daclatasvir, asunaprevir, beclabuvir and sofosbuvir (FOURward study). Liver Int. 2017 Jun;37(6):836-842. doi: 10.1111/liv.13335. Epub 2017 Feb 2. PMID 27943563
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 participants enrolled in the study, 28 were randomized. Of the 7 not randomized, 1 participant withdrew consent and 6 no longer met study criteria
Groups:
- 4 Weeks DCV 3DAA + SOF: Oral dose of a fixed dose combination regimen administered as 1 tablet BID comprising of 30 mg daclatasvir, 200 mg asunaprevir, and 75 mg beclabuvir (referred to as DCV 3DAA), plus sofosbuvir 400 mg 1 tablet daily for 4 weeks (treatment period). Thereafter, participants entered a follow-up period of 24 weeks after completion of study treatment or upon early discontinuation of treatment.
- 6 Weeks DCV 3DAA + SOF: Oral dose of a fixed dose combination regimen administered as 1 tablet BID comprising of 30 mg daclatasvir, 200 mg asunaprevir, and 75 mg beclabuvir, plus sofosbuvir 400 mg 1 tablet daily for 6 weeks (treatment period). Thereafter, participants entered a follow-up period of 24 weeks after completion of study treatment or upon early discontinuation of treatment.
Period: Treatment Period
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Follow-up Period
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Started | 14 | 14
Completed | 4 | 8
Not Completed | 10 | 6
Not completed — Lack of Efficacy | 10 | 6

BASELINE CHARACTERISTICS:
Population: All treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Full Range); unit: years] | 58.0 [21 to 64] | 59.0 [31 to 64] | 58.5 [21 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 (SVR12)
Description: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) < lower limit of quantitation (LLOQ) target detected (TD) or not detected (TND) at post-treatment follow-up Week 12. Imputed SVR12 was based on Next Value Carried Backwards approach.
Time Frame: 12 Weeks after treatment discontinuation (Follow-up Week 12)
Population: It included treated participants (randomized participants) who received at least 1 dose of study therapy (DCV 3DAA or SOF).
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Number analyzed (Participants) | 14 | 14
Percentage of participants | 28.6 [13.1 to 49.2] | 57.1 [36.9 to 75.7]

2. Secondary Outcome: Percentage of Participants With End of Treatment Response (EOTR)
Description: EOTR was defined as HCV RNA less than the lower limit of quantitation, target detected or not detected at end of treatment.
Time Frame: End of the treatment
Population: All treated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Number analyzed (Participants) | 14 | 14
Percentage of participants | 92.9 [66.1 to 99.8] | 100.0 [76.8 to 100.0]

3. Primary Outcome: Number of Participants With Deaths, Serious Adverse Events (SAEs) and AEs Leading to Discontinuation From Treatment
Description: SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/ birth defect.
Time Frame: From signature of the informed consent until 4 weeks after last treatment administration.(Approximately 17 months)
Population: Safety population included participants who received at least 1 dose of study therapy (DCV 3DAA or SOF).
Measure: Count of Participants; unit: Participants
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Number analyzed (Participants) | 14 | 14
Participants
  Death | 0 | 0
  Serious Adverse Events | 1 | 0
  AEs Leading to Discontinuation | 0 | 0

4. Primary Outcome: Number of Participants With Selected Grade 3/4 Laboratory Abnormalities
Description: Grade 3/4 laboratory abnormalities (hematology, electrolyte, lipase, liver function, metabolic, renal function, urinalysis). The Week 24 data set was used to evaluate the Week-24 on-treatment safety. The cumulative data set was used to evaluate the safety while on treatment. Common Terminology Criteria for Adverse Events v3.0 (CTCAE) Grades:1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death.
Time Frame: From signature of the informed consent until 4 weeks after last treatment administration.(Approximately 17 months)
Population: Safety analysis population included participants who received at least 1 dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

5. Secondary Outcome: Percentage of Participants Who Achieved HCV RNA <LLOQ TD/TND
Description: Percentage of Participants with hepatitis C virus(HCV) ribonucleic acid (RNA) < lower limit of quantitation (LLOQ), target detected (TD) or target not detected (TND) were presented at treatment Weeks 1, 2, 4, 6, and follow-up Weeks 2 (SVR2), 4 (SVR4), 12 (SVR12) and 24 (SVR24).
Time Frame: Treatment Weeks 1, 2, 4 and 6; post-treatment Weeks 2 (SVR2), 4 (SVR4), 12 (SVR12) and 24 (SVR24)
Population: It included modified Intent-to-treat treated population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Number analyzed (Participants) | 14 | 14
Percentage of Participants
  Week 1 | 35.7 [12.8 to 64.9] | 71.4 [41.9 to 91.6]
  Week 2 | 78.6 [49.2 to 95.3] | 100.0 [76.8 to 100.0]
  Week 4 | 100.0 [76.8 to 100.0] | 100.0 [76.8 to 100.0]
  Week 6 | NA [NA to NA] — NA signifies data was not estimable due to lesser number of events. | 100.0 [76.8 to 100.0]
  Follow-Up Week 2 | 78.6 [49.2 to 95.3] | 100.0 [76.8 to 100.0]
  Follow-Up Week 4 | 42.9 [17.7 to 71.1] | 78.6 [49.2 to 95.3]
  Follow-Up Week 12 | 28.6 [8.4 to 58.1] | 57.1 [28.9 to 82.3]
  Follow-Up Week 24 | 28.6 [8.4 to 58.1] | 57.1 [28.9 to 82.3]

6. Secondary Outcome: Percentage of Participants Who Achieved HCV RNA < LLOQ TND
Description: Percentage of Participants with hepatitis C virus(HCV) ribonucleic acid (RNA) < lower limit of quantitation (LLOQ), target not detected (TND) were presented at treatment Weeks 1, 2, 4, 6, and follow-up Weeks 2 (SVR2), 4 (SVR4), and 24 (SVR24).
Time Frame: Treatment Weeks 1, 2, 4 and 6; post-treatment Weeks 2, 4, 12 and 24
Population: It included modified ITT treated population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Number analyzed (Participants) | 14 | 14
Percentage of participants
  Week 1 | 21.4 [4.7 to 50.8] | 7.1 [0.2 to 33.9]
  Week 2 | 42.9 [17.7 to 71.1] | 64.3 [35.1 to 87.2]
  Week 4 | 92.9 [66.1 to 99.8] | 100.0 [76.8 to 100.0]
  Week 6 | NA [NA to NA] — NA signifies data was not reported due to lesser number of events. | 100.0 [76.8 to 100.0]
  Follow-Up Week 2 | 71.4 [41.9 to 91.6] | 92.9 [66.1 to 99.8]
  Follow-Up Week 4 | 42.9 [17.7 to 71.1] | 71.4 [41.9 to 91.6]
  Follow-Up Week 12 | 28.6 [8.4 to 58.1] | 57.1 [28.9 to 82.3]
  Follow-Up Week 24 | 28.6 [8.4 to 58.1] | 57.1 [28.9 to 82.3]

7. Secondary Outcome: Percentage of Participants Who Achieved SVR12 Associated With HCV Geno Subtype 1a vs 1b
Description: Percentage of Participants who Achieved SVR12 Associated with HCV geno subtype 1a or 1b
Time Frame: Post-treatment Week 12
Population: All included treated participants. Here n' signifies number of participants analysed for specific category.
Measure: Number; unit: Percentage of Participants
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Number analyzed (Participants) | 14 | 14
Percentage of Participants
  Genotype 1a: number analyzed (Participants) | 11 | 11
  Genotype 1a | 27.3 | 54.5
  Genotype 1b: number analyzed (Participants) | 3 | 3
  Genotype 1b | 33.3 | 66.7

8. Secondary Outcome: Percentage of Participants Who Achieved SVR12 Associated With Interleukin-28B (IL28B) rs12979860 SNP Status (CC Genotype or Non-CC Genotype)
Description: Percentage of Participants who Achieved SVR12 Associated with IL28B rs12979860 Single Nucleotide Polymorphisms (SNP) status (CC genotype or non CC genotype) were reported.
Time Frame: Post-treatment Week 12
Population: All included treated participants. Here, n' signifies number of participants analysed for specific category.
Measure: Number; unit: Percentage of Participants
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
Number analyzed (Participants) | 14 | 14
Percentage of Participants
  CC genotype: number analyzed (Participants) | 5 | 6
  CC genotype | 40.0 | 66.7
  Non-CC Genotype: number analyzed (Participants) | 9 | 8
  Non-CC Genotype | 22.2 | 50.0

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent until 4 weeks after last treatment administration.(Approximately 17 months)
Arm/Group | 4 Weeks DCV 3DAA + SOF | 6 Weeks DCV 3DAA + SOF
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/14 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 Weeks DCV 3DAA + SOF (N=14) | 6 Weeks DCV 3DAA + SOF (N=14)
Overdose (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4 Weeks DCV 3DAA + SOF (N=14) | 6 Weeks DCV 3DAA + SOF (N=14)
FATIGUE (General disorders) | 3 | 4
CHEST DISCOMFORT (General disorders) | 0 | 1
CHILLS (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 2 | 3
DIZZINESS (Nervous system disorders) | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1
ORAL HERPES (Infections and infestations) | 0 | 1
SINUSITIS (Infections and infestations) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 1 | 1
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
INSOMNIA (Psychiatric disorders) | 0 | 2
AFFECT LABILITY (Psychiatric disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0
FLUSHING (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period <=60 days from submitting for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.